CLINICAL TRIAL: NCT02754180
Title: Adjuvant Gemcitabine Versus Gemcitabine With Chemoradiation in Pancreatic Adenocarcinoma With R1 Resection and/or Positive Lymph Nodes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, YueJuan Cheng, MD, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-1015
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Neoplasms
Keywords: adjuvant; pancreatic cancer; R1 resection; positive lymph nodes
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Drug Therapy; titanium silicide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy (Active Comparator): gemcitabine 1g/m2 iv d1, 8, 15, q4wks. 6 cycles.
  Interventions: Drug: Gemcitabine
- chemotherapy with chemoradiation (Experimental): gemcitabine 1g/m2 iv d1, 8, 15, q4wks. 6 cycles. Followed by TS-1 based chemoradiation. TS-1 40mg/m2 bid, 5 days/week, with radiation.
  Interventions: Drug: Gemcitabine; Radiation: TS-1 with radiation

INTERVENTIONS:
Drug: Gemcitabine — gemcitabine 1g/m2 iv d1, 8, 15, q4wks. 6 cycles
  Other Names: chemotherapy
Radiation: TS-1 with radiation — gemcitabine 1g/m2 iv d1, 8, 15, q4wks. 6 cycles. Followed by TS-1 based chemoradiation. TS-1 40mg/m2 bid, 5 days/week, with radiation.
  Arms: chemotherapy with chemoradiation

SUMMARY:
Adjuvant Gemcitabine Versus Gemcitabine With Chemoradiation in Pancreatic Adenocarcinoma With R1 Resection and/or Positive Lymph Nodes after curative resection.

DETAILED DESCRIPTION:
Adjuvant Gemcitabine Versus Gemcitabine With TS-1 based Chemoradiation in Pancreatic Adenocarcinoma With R1 Resection and/or Positive Lymph Nodes after curative resection: a randomized phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed resected ductal pancreatic adenocarcinoma with R1 resection and/or positive lymph nodes.
* Subject should start treatment no later than 10 weeks postsurgery.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Acceptable hematology parameters:

  * Absolute neutrophil count ≥1500 cell/mm3
  * Platelet count ≥100,000/mm3
  * Hemoglobin (Hgb) ≥8.0 g/dL
* Acceptable blood chemistry levels:

  * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤2.5 × upper limit of normal range (ULN)
  * Total bilirubin ≤ 2.5 x upper Limit of Normal (ULN)
  * Serum creatinine within upper limits of normal.
* Cancer antigen (CA)19-9 ≤ 2.5 x upper Limit of Normal (ULN) assessed within 14 days of randomization.
* No disease recurrence or metastases detected on CT/MRI assessed within 30 days of randomization.
* Signed informed consent.

Exclusion Criteria:

* R2 resection or presence of metastatic disease.
* Prior neo-adjuvant treatment or radiation therapy for pancreatic adenocarcinoma.
* Any other malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, bladder, or nonmelanomatous skin cancer.
* Active, uncontrolled infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the 6 months of study registration
  * Uncontrolled hypertension, diabetes or arrhythmia.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization.
* Not able to take medicine orally.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of randomization until the date of first documented disease recurrence or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 36 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | from randomization to 1 month after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No